CLINICAL TRIAL: NCT03441633
Title: APIXABAN DRUG UTILIZATION STUDY IN STROKE PREVENTION IN ATRIAL FIBRILLATION (SPAF)
Acronym: SPAF
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661076; SPAF (Other: Alias Study Number)
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Results first posted 2019-04-19 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; apixaban; stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — apixaban; Dabigatran; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1. Apixaban: Patients who are on treatment with apixaban.
  1a. patients who have initiated with apixaban as treatment naïve (no prior prescription of VKA previous to the 12 months before index date).
  1b. patients who previously have been treated with VKA in the 12 months before index date.
  Interventions: Drug: apixaban
- Group 2. VKA: Patients who are on treatment with VKA.
  2a. patients who have initiated with VKA as treatment naïve (no prior prescription of VKA previous to the 12 months before index date).
  2b. patients who previously have been treated with VKA in the 12 months before index date.
  Interventions: Drug: VKA
- Group 3. Dabigatran: Patients who are on treatment with dabigatran.
  3a. patients who have initiated with dabigatran as treatment naïve (no prior prescription of VKA previous to the 12 months before index date).
  3b. patients who previously have been treated with VKA in the 12 months before index date.
  Interventions: Drug: dabigatran
- Group 4. Rivaroxaban: Patients who are on treatment with rivaroxaban.
  4a. patients who have initiated with rivaroxaban as treatment naïve (no prior prescription of VKA previous to the 12 months before index date).
  4b. patients who previously have been treated with VKA in the 12 months before index date.
  Interventions: Drug: rivaroxaban

INTERVENTIONS:
Drug: apixaban — current or new medication
  Groups: Group 1. Apixaban
Drug: dabigatran — current or new medication
  Groups: Group 3. Dabigatran
Drug: VKA — current or new medication
  Groups: Group 2. VKA
Drug: rivaroxaban — current or new medication
  Groups: Group 4. Rivaroxaban

SUMMARY:
Apixaban is a direct anticoagulant, which inhibits the factor Xa. Its clinical efficiency in prevention of stroke and systemic embolism in adult patients with NVAF (non/valvular atrial fibrillation) was demonstrated as well as has shown better safety profile compared with warfarin. A Drug Utilization study will evaluate whether this drug has been used in accordance with the approved indication and recommendations described in the summary of product characteristics (SmPC) and estimate possible misuse or overuse apixaban.

DETAILED DESCRIPTION:
The primary research question is to evaluate the apixaban utilization according to the approved SPAF indication and recommendations by EMA.

In addition a comparison with a cohort of NVAF patients treated with VKA, dabigatran and rivaroxaban for the SPAF indication will also be performed.

Objective 1: To characterize patients using apixaban according to demographics, comorbidity, risk of thromboembolic events (CHADS2 and CHA2DS2-Vasc scores), risk of bleeding events (HAS-BLED score), comedications and compare it with the profile of patients treated with VKA, dabigatran and rivaroxaban.

Objective 2: Describe the level of appropriate usage according to the posology recommended in the apixaban SmPC.

Objective 3: Describe the potential interactions with other drugs prescribed concomintatly according with the SmPC recommendations.

Objective 4: Estimate the level of apixaban adherence by the medication possession ratio (MPR) and discontinuation rates and compare it with VKA, dabigatran and rivaroxaban cohort.

Objective 5: To analyze INR (International Normalized Ratio) values during the last 12 months and to obtain TTR (Time in Therapeutic Range) values in patients previously treated with VKA, and during the whole study period for those in the cohort treated with VKA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients more than 18 years-old.
2. Patients diagnosed with NVAF registered in primary care according to ICD-10.
3. Patients initiating apixaban (naïve or VKA experienced), VKA (naïve or VKA experienced), dabigatran or rivaroxaban for the SPAF indication.
4. Continuous enrolment in the 12 months pre-index.

Exclusion Criteria:

1. Patients with valvular heart disease (ICD 10: I05.0-I05.09, I08.0-I08.9) including patients with mitral prosthetic valves.
2. Lost to follow-up (e.g. transfer to primary care center non-ICS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SIDIAP currently collects information from 274 primary health care centers, including more than 5.8 million patients, about 80 % of the Catalonia population, or more than 10 % of the Spanish population covered by the Catalan Institute of Health.
  The study population for these cohorts includes all eligible subjects from the source population with a first -recorded prescription of apixaban VKA, dabigatran or rivaroxaban for the SPAF indication, registered in SIDIAP database and diagnosis of NVAF for study period.
Sampling Method: Probability Sample
Enrollment: 51690 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- IDIAP Jordi Gol, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0661076&StudyName=APIXABAN+DRUG+UTILIZATION+STUDY+IN+STROKE+PREVENTION+IN+ATRIAL+FIBRILLATION+%28SPAF%29

RESULTS

PARTICIPANT FLOW:
Groups:
- Apixaban: Naive: Participants who were treated with apixaban without prior prescription of vitamin K antagonists (VKA) (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban during 12 months before start date (when the participant took the drug for the first time). The dose and frequency of drug was as per treating physician.
- Apixaban: Non Naive: Participants who were treated with apixaban with prior prescription of VKA (warfarin or acenocoumarol), dabigatran or rivaroxaban in the 12 months before start date. The dose and frequency of drug was as per treating physician.
- Acenocoumarol: Naive: Participants who were treated with acenocoumarol without prior prescription of VKA (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban during 12 months before start date. The dose and frequency of drug was as per treating physician.
- Acenocoumarol: Non-Naive: Participants who were treated with acenocoumarol with prior prescription of different VKA (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban in the 12 months before start date. The dose and frequency of drug was as per treating physician.
- Warfarin: Naive: Participants who were treated with warfarin without prior prescription of VKA (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban during 12 months before start date. The dose and frequency of drug was as per treating physician.
- Warfarin: Non-Naive: Participants who were treated with warfarin with prior prescription of different VKA (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban in the 12 months before start date. The dose and frequency of drug was as per treating physician.
- Dabigatran: Naive: Participants who were treated with dabigatran without prior prescription of VKA (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban during 12 months before start date. The dose and frequency of drug was as per treating physician.
- Dabigatran: Non-Naive: Participants who were treated with dabigatran with prior prescription of VKA (warfarin or acenocoumarol), apixaban or rivaroxaban in the 12 months before start date. The dose and frequency of drug was as per treating physician.
- Rivaroxaban: Naive: Participants who were treated with rivaroxaban without prior prescription of VKA (warfarin or acenocoumarol), apixaban, dabigatran or rivaroxaban during 12 months before start date. The dose and frequency of drug was as per treating physician.
- Rivaroxaban: Non-Naive: Participants who were treated with rivaroxaban with prior prescription of VKA (warfarin or acenocoumarol), apixaban and dabigatran in the 12 months before start date. The dose and frequency of drug was as per treating physician.
Period: Overall Study
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Started | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Completed | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study population included all participants with a first-recorded prescription of apixaban, VKA, dabigatran or rivaroxaban for stroke prevention in atrial fibrillation(SPAF) registered in information system for the improvement of research in primary care(SIDIAP) database during the study and diagnosed with non-valvular atrial fibrillation(NVAF).
Groups:
- Warfarin: Non Naive: Participants who were treated with warfarin with prior prescription of different VKA, apixaban, dabigatran or rivaroxaban in the 12 months before start date. The dose and frequency of drug was as per treating physician.
- Total: Total of all reporting groups
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive | Total
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562 | 51690
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (11.1) | 78.1 (8.7) | 73.5 (12.3) | 74.6 (10.7) | 69.7 (13.4) | 74.9 (12.9) | 69.9 (12.3) | 76.5 (9.5) | 69.3 (13.2) | 76.4 (10.5) | 72.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2661 | 751 | 15531 | 94 | 979 | 205 | 1399 | 479 | 2649 | 811 | 25559
  Male | 2051 | 672 | 16681 | 98 | 1307 | 158 | 1456 | 474 | 2483 | 751 | 26131
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Their Sociodemographic Characteristics: Smoking Habit
Description: Socio-demographics were characteristics of a population. One of the socio-demographics characteristics included smoking habit.
Time Frame: Day 1
Population: Study population included all participants with a first-recorded prescription of apixaban, VKA, dabigatran or rivaroxaban for SPAF registered in SIDIAP database during the study and diagnosed with NVAF.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Participants
  Missing | 207 | 23 | 1844 | 7 | 112 | 14 | 225 | 23 | 354 | 38
  Non-smoker | 3104 | 946 | 19440 | 119 | 1166 | 234 | 1684 | 623 | 3079 | 1030
  Ex-smoker | 459 | 83 | 3676 | 16 | 320 | 26 | 355 | 72 | 608 | 102
  Smoker | 942 | 371 | 7252 | 50 | 688 | 89 | 591 | 235 | 1091 | 392
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Non-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.68 to 0.82]
Statistical Analysis 2: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Ex-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.32, 95% CI 2-sided [1.14 to 1.52]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.93 to 1.17]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Non-smoker); Test type: Superiority; p = 0.755, Chi-squared; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.80 to 1.13]
Statistical Analysis 5: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Ex-smoker); Test type: Superiority; p = 0.426, Chi-squared; Odds Ratio (OR) = 1.32, 95% CI 2-sided [0.95 to 1.83]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Smoker); Test type: Superiority; p = 0.930, Chi-squared; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.77 to 1.12]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Non-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.72 to 0.84]
Statistical Analysis 8: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Ex-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.10 to 1.42]
Statistical Analysis 9: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.98 to 1.19]
Statistical Analysis 10: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Non-smoker); Test type: Superiority; p = 0.755, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.84 to 1.14]
Statistical Analysis 11: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Ex-smoker); Test type: Superiority; p = 0.426, Chi-squared; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.84 to 1.52]
Statistical Analysis 12: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Smoker); Test type: Superiority; p = 0.930, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.81 to 1.12]
Statistical Analysis 13: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Non-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.74 to 0.84]
Statistical Analysis 14: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Ex-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.19, 95% CI 2-sided [1.08 to 1.32]
Statistical Analysis 15: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.16, 95% CI 2-sided [1.08 to 1.26]
Statistical Analysis 16: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Non-smoker); Test type: Superiority; p = 0.755, Chi-squared; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.60 to 1.13]
Statistical Analysis 17: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Ex-smoker); Test type: Superiority; p = 0.426, Chi-squared; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.82 to 2.52]
Statistical Analysis 18: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Smoker); Test type: Superiority; p = 0.930, Chi-squared; Odds Ratio (OR) = 1.00, 95% CI 2-sided [0.70 to 1.40]
Statistical Analysis 19: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Non-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.54, 95% CI 2-sided [0.49 to 0.60]
Statistical Analysis 20: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Ex-smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.29 to 1.76]
Statistical Analysis 21: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Smoker); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.54 to 1.93]
Statistical Analysis 22: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Non-smoker); Test type: Superiority; p = 0.755, Chi-squared; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.72 to 1.17]
Statistical Analysis 23: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Ex-smoker); Test type: Superiority; p = 0.426, Chi-squared; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.78 to 1.95]
Statistical Analysis 24: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in naive participants (Smoker); Test type: Superiority; p = 0.930, Chi-squared; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.70 to 1.20]

2. Primary Outcome: Number of Participants by Their Sociodemographic Characteristics: Alcoholic Habit
Description: Socio-demographics were characteristics of a population. One of the socio-demographics characteristics included alcoholic habit.
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Participants
  Missing | 2162 | 353 | 11299 | 40 | 839 | 91 | 1263 | 211 | 2475 | 366
  No intake | 1749 | 810 | 14337 | 111 | 984 | 212 | 1054 | 550 | 1696 | 923
  Moderate intake | 765 | 247 | 6241 | 39 | 447 | 58 | 505 | 187 | 915 | 255
  Risk consumption | 36 | 13 | 335 | 2 | 16 | 2 | 33 | 5 | 46 | 18
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (No intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.90 to 1.09]
Statistical Analysis 2: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Moderate intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.98 to 1.25]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Risk consumption); Test type: Superiority; p = 0.164, Chi-squared; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.94 to 2.45]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (No intake); Test type: Superiority; p = 0.826, Chi-squared; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.87 to 1.22]
Statistical Analysis 5: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Moderate intake); Test type: Superiority; p = 0.190, Chi-squared; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.94 to 1.43]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Risk consumption); Test type: Superiority; p = 0.526, Chi-squared; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.18 to 1.57]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (No intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.77 to 0.91]
Statistical Analysis 8: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Moderate intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.12, 95% CI 2-sided [1.01 to 1.24]
Statistical Analysis 9: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Risk consumption); Test type: Superiority; p = 0.164, Chi-squared; Odds Ratio (OR) = 1.17, 95% CI 2-sided [0.76 to 1.83]
Statistical Analysis 10: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (No intake); Test type: Superiority; p = 0.826, Chi-squared; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.95 to 1.26]
Statistical Analysis 11: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Moderate intake); Test type: Superiority; p = 0.190, Chi-squared; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.77 to 1.13]
Statistical Analysis 12: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Risk consumption); Test type: Superiority; p = 0.526, Chi-squared; Odds Ratio (OR) = 1.26, 95% CI 2-sided [0.62 to 2.65]
Statistical Analysis 13: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (No intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.28 to 1.45]
Statistical Analysis 14: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Moderate intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.24, 95% CI 2-sided [1.14 to 1.35]
Statistical Analysis 15: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Risk consumption); Test type: Superiority; p = 0.164, Chi-squared; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.98 to 1.95]
Statistical Analysis 16: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (No intake); Test type: Superiority; p = 0.826, Chi-squared; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.76 to 1.41]
Statistical Analysis 17: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Moderate intake); Test type: Superiority; p = 0.190, Chi-squared; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.82 to 1.76]
Statistical Analysis 18: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Risk consumption); Test type: Superiority; p = 0.526, Chi-squared; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.17 to 4.50]
Statistical Analysis 19: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (No intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.28, 95% CI 2-sided [1.16 to 1.42]
Statistical Analysis 20: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Moderate intake); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.25, 95% CI 2-sided [1.10 to 1.43]
Statistical Analysis 21: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Risk consumption); Test type: Superiority; p = 0.164, Chi-squared; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.49 to 1.64]
Statistical Analysis 22: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (No intake); Test type: Superiority; p = 0.826, Chi-squared; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.84 to 1.34]
Statistical Analysis 23: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Moderate intake); Test type: Superiority; p = 0.190, Chi-squared; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.66 to 1.23]
Statistical Analysis 24: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Risk consumption); Test type: Superiority; p = 0.526, Chi-squared; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.09 to 2.36]

3. Primary Outcome: Number of Participants by Their Sociodemographic Characteristics: MEDEA
Description: Socio-demographics were characteristics of a population. One of the socio-demographics characteristics included MEDEA. MEDEA was a deprivation index that was associated with overall mortality in urban areas. It included factors like job, education, housing conditions and single parent homes. The MEDEA index was categorized in quintiles for urban areas, with quintile 1 corresponding to the least deprived population and quintile 5, the most deprived.
Time Frame: Day 1
Population: Study population included all participants with a first-recorded prescription of apixaban, VKA, dabigatran or rivaroxaban for SPAF registered in SIDIAP database during the study and diagnosed with NVAF. Here, "Overall Number of Participants Analyzed (N)" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4027 | 1210 | 25477 | 154 | 2163 | 322 | 2393 | 789 | 4430 | 1389
Participants
  Missing - Urban area | 190 | 90 | 1754 | 16 | 120 | 28 | 110 | 57 | 230 | 145
  Quintile 1 - Urban area | 716 | 224 | 4735 | 31 | 149 | 73 | 558 | 156 | 973 | 230
  Quintile 2 - Urban area | 754 | 216 | 4753 | 25 | 315 | 73 | 461 | 148 | 803 | 234
  Quintile 3 - Urban area | 825 | 256 | 4801 | 27 | 606 | 52 | 447 | 137 | 904 | 230
  Quintile 4 - Urban area | 807 | 231 | 4744 | 28 | 635 | 55 | 429 | 152 | 837 | 300
  Quintile 5 - Urban area | 735 | 193 | 4690 | 27 | 338 | 41 | 388 | 139 | 683 | 250
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.36, 95% CI 2-sided [1.20 to 1.53]
Statistical Analysis 2: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.014, Chi-squared; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.89 to 1.15]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.77 to 0.99]
Statistical Analysis 4: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.75 to 0.97]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.013, Chi-squared; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.74 to 0.97]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.157, Chi-squared; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.84 to 1.31]
Statistical Analysis 7: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.124, Chi-squared; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.82 to 1.29]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.062, Chi-squared; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.61 to 0.96]
Statistical Analysis 9: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.079, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.78 to 1.22]
Statistical Analysis 10: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.140, Chi-squared; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.86 to 1.38]
Statistical Analysis 11: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.31, 95% CI 2-sided [1.17 to 1.45]
Statistical Analysis 12: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.014, Chi-squared; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.87 to 1.09]
Statistical Analysis 13: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.91 to 1.12]
Statistical Analysis 14: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.85 to 1.05]
Statistical Analysis 15: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.013, Chi-squared; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.74 to 0.93]
Statistical Analysis 16: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.157, Chi-squared; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.76 to 1.13]
Statistical Analysis 17: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.124, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.81 to 1.20]
Statistical Analysis 18: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.062, Chi-squared; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.65 to 0.96]
Statistical Analysis 19: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.079, Chi-squared; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.02 to 1.48]
Statistical Analysis 20: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.140, Chi-squared; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.99 to 1.49]
Statistical Analysis 21: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.88 to 1.05]
Statistical Analysis 22: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.014, Chi-squared; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.84 to 0.99]
Statistical Analysis 23: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.76 to 0.90]
Statistical Analysis 24: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.77 to 0.91]
Statistical Analysis 25: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.013, Chi-squared; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.85 to 1.00]
Statistical Analysis 26: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.157, Chi-squared; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.68 to 1.54]
Statistical Analysis 27: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.124, Chi-squared; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.53 to 1.29]
Statistical Analysis 28: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.062, Chi-squared; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.48 to 1.13]
Statistical Analysis 29: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.079, Chi-squared; Odds Ratio (OR) = 0.88, 95% CI 2-sided [0.57 to 1.33]
Statistical Analysis 30: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.140, Chi-squared; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.67 to 1.59]
Statistical Analysis 31: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.32 to 0.47]
Statistical Analysis 32: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.014, Chi-squared; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.73 to 0.97]
Statistical Analysis 33: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.70, 95% CI 2-sided [1.51 to 1.91]
Statistical Analysis 34: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.86, 95% CI 2-sided [1.65 to 2.10]
Statistical Analysis 35: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.013, Chi-squared; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.82 to 1.08]
Statistical Analysis 36: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Quintile 1 - Urban area); Test type: Superiority; p = 0.157, Chi-squared; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.00 to 1.80]
Statistical Analysis 37: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Quintile 2 - Urban area); Test type: Superiority; p = 0.124, Chi-squared; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.04 to 1.88]
Statistical Analysis 38: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Quintile 3 - Urban area); Test type: Superiority; p = 0.062, Chi-squared; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.55 to 1.05]
Statistical Analysis 39: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Quintile 4 - Urban area); Test type: Superiority; p = 0.079, Chi-squared; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.67 to 1.26]
Statistical Analysis 40: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Quintile 5 - Urban area); Test type: Superiority; p = 0.140, Chi-squared; Odds Ratio (OR) = 0.81, 95% CI 2-sided [0.56 to 1.15]

4. Primary Outcome: Number of Participants by Their Sociodemographic Characteristics: Body Mass Index (BMI)
Description: Socio-demographics were characteristics of a population. One of the socio-demographics characteristics included BMI. BMI was defined as an index for assessing overweight and underweight and was obtained by dividing body weight in kilograms (kg) by height in meters squared (m^2).
Time Frame: Day 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Participants
  Missing | 1424 | 261 | 6898 | 34 | 509 | 87 | 960 | 178 | 1746 | 311
  18.5 - 25 kg per m^2 (Normal) | 423 | 253 | 4471 | 30 | 295 | 78 | 272 | 144 | 464 | 271
  Less than (<) 18.5 kg per m^2 (Underweight) | 12 | 6 | 141 | 0 | 6 | 2 | 10 | 8 | 16 | 0
  25 - 30 kg per m^2 (Overweight) | 1229 | 493 | 10074 | 68 | 712 | 119 | 735 | 306 | 1289 | 482
  Greater than (>) 30 kg per m^2 (Obese) | 1624 | 410 | 10628 | 60 | 764 | 77 | 878 | 317 | 1617 | 498
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.91 to 1.25]
Statistical Analysis 2: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.202, Chi-squared; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.58 to 3.23]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.88 to 1.09]
Statistical Analysis 4: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.003, Chi-squared; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.76 to 0.93]
Statistical Analysis 5: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.083, Chi-squared; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.66 to 1.03]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.011, Chi-squared; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.68 to 6.18]
Statistical Analysis 7: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.227, Chi-squared; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.75 to 1.06]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.23, 95% CI 2-sided [1.03 to 1.47]
Statistical Analysis 9: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.88 to 1.16]
Statistical Analysis 10: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.202, Chi-squared; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.58 to 2.66]
Statistical Analysis 11: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.87 to 1.04]
Statistical Analysis 12: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.003, Chi-squared; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.80 to 0.95]
Statistical Analysis 13: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.083, Chi-squared; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.80 to 1.17]
Statistical Analysis 14: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.011, Chi-squared; Odds Ratio (OR) = 0.06, 95% CI 2-sided [0.02 to 1.05]
Statistical Analysis 15: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.227, Chi-squared; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.72 to 0.98]
Statistical Analysis 16: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.99 to 1.35]
Statistical Analysis 17: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.63, 95% CI 2-sided [1.47 to 1.82]
Statistical Analysis 18: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.202, Chi-squared; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.98 to 3.25]
Statistical Analysis 19: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocoumarol vs. Apixaban in naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.29, 95% CI 2-sided [1.20 to 1.38]
Statistical Analysis 20: Comparison: Apixaban: Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.003, Chi-squared; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.88 to 1.00]
Statistical Analysis 21: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.083, Chi-squared; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.56 to 1.28]
Statistical Analysis 22: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.011, Chi-squared; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.13 to 8.58]
Statistical Analysis 23: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.227, Chi-squared; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.75 to 1.42]
Statistical Analysis 24: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocoumarol vs. Apixaban in non-naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.81 to 1.55]
Statistical Analysis 25: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.50, 95% CI 2-sided [1.28 to 1.76]
Statistical Analysis 26: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.202, Chi-squared; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.36 to 2.73]
Statistical Analysis 27: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.28, 95% CI 2-sided [1.15 to 1.43]
Statistical Analysis 28: Comparison: Apixaban: Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.003, Chi-squared; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.86 to 1.06]
Statistical Analysis 29: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (18.5 - 25 kg per m^2 Normal); Test type: Superiority; p = 0.083, Chi-squared; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.95 to 1.68]
Statistical Analysis 30: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (<18.5 kg per m^2 Underweight); Test type: Superiority; p = 0.011, Chi-squared; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.18 to 6.21]
Statistical Analysis 31: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (25 - 30 kg per m^2 Overweight); Test type: Superiority; p = 0.227, Chi-squared; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.72 to 1.17]
Statistical Analysis 32: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (>30 kg per m^2 Obese); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.50 to 0.87]

5. Primary Outcome: Number of Participants by Comorbidity
Description: Comorbidity was defined as the presence of one or more additional diseases or disorders co-occurring with (that is, concomitant or concurrent with) a primary disease or disorder.
Time Frame: Up to 12 months after date of first prescription
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Participants | 3695 | 1316 | 26450 | 173 | 1819 | 318 | 2030 | 870 | 3731 | 1417
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants; Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.61 to 0.75]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.052, Chi-squared; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.63 to 1.15]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants; Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.67 to 0.80]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.052, Chi-squared; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.61 to 1.03]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants; Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.17 to 1.36]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.052, Chi-squared; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.45 to 1.27]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants; Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.95 to 1.21]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.052, Chi-squared; Odds Ratio (OR) = 0.57, 95% CI 2-sided [0.40 to 0.84]

6. Primary Outcome: Risk of Bleeding Events: HAS-BLED Score
Description: Risk of bleeding events was assessed by using HAS-BLED score. HAS-BLED was a scoring system that was developed to assess 1 year risk of occurrence of major hemorrhage. HAS-BLED score was assessed by combining score of 9 risk factors: hypertension history, renal disease, liver disease, stroke history, prior major bleeding or predisposition to bleeding, labile international normalized ratio (INR), age >65 years, medication usage predisposing to bleeding and alcohol or drug usage history. The total score ranged from 0 to 9 where 0 = low risk of bleed per 100 participants-year and >3 = high risk of bleed per 100 participants-year.
Time Frame: Up to 12 months prior to enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: bleed per 100 participants-year
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
bleed per 100 participants-year | 1.7 (1.0) | 2.7 (1.1) | 2.2 (1.1) | 2.5 (1.0) | 1.9 (1.1) | 2.4 (1.2) | 1.5 (1.0) | 2.6 (1.0) | 1.6 (1.0) | 2.6 (1.1)
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (HAS - BLED); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-0.26 to -0.17]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (HAS - BLED); Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.18 to -0.01]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (HAS - BLED); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.23 to -0.15]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (HAS - BLED); Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.19 to -0.04]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (HAS - BLED); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [0.47 to 0.53]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (HAS - BLED); Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.32 to -0.02]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (HAS - BLED); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [0.12 to 0.23]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (HAS - BLED); Test type: Superiority; p = 0.001, ANOVA; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-0.37 to -0.10]

7. Primary Outcome: Risk of Thromboembolic Events: CHADS2 Score
Description: Thromboembolic events were defined as an embolic stroke that occurred when a blood clot that formed elsewhere in the body breaks loose and travels to the brain via bloodstream. Risk of thromboembolic events was calculated using CHADS2 score. CHADS2 score was assessed by combining score of 5 risk factors (congestive heart failure history, hypertension history, age >=75 years, diabetes mellitus history and stroke/transient ischemic attack symptoms previously). Total CHADS2 score ranged from 0-6 where 0 =low risk and 6 =high risk of stroke.
Time Frame: Up to 12 months prior to enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: stroke risk per year
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
stroke risk per year | 1.7 (1.3) | 2.8 (1.4) | 1.9 (1.3) | 2.3 (1.3) | 1.8 (1.3) | 2.5 (1.5) | 1.5 (1.3) | 2.6 (1.4) | 1.5 (1.2) | 2.6 (1.4)
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.24 to -0.12]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.35 to -0.12]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.28 to -0.18]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.31 to -0.11]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [0.17 to 0.25]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-0.70 to -0.30]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.01 to 0.14]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (CHADS2); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.54 to -0.20]

8. Primary Outcome: Risk of Thromboembolic Events: CHA2DS2Vasc Score
Description: Thromboembolic events were defined as an embolic stroke that occurred when a blood clot that formed elsewhere in the body breaks loose and travels to the brain via bloodstream. Risk of thromboembolic events was calculated using CHA2DS2Vasc score. CHA2DS2Vasc score was assessed by combining score of 8 risk factors (female, >=65 and <75 years, congestive heart failure history, hypertension history, diabetes mellitus history, vascular disease history, age >=75 years and stroke/TIA symptoms previously). Total CHA2DS2Vasc score ranged from 0-9 where 0=low risk and 9=high risk of stroke.
Time Frame: Up to 12 months prior to enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: stroke risk per year
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
stroke risk per year | 3.0 (1.7) | 4.4 (1.6) | 3.2 (1.7) | 3.7 (1.6) | 2.9 (1.8) | 3.9 (1.9) | 2.7 (1.8) | 4.0 (1.7) | 2.7 (1.7) | 4.1 (1.7)
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.42 to -0.26]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-0.46 to -0.19]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.38, 95% CI 2-sided [-0.45 to -0.32]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.39 to -0.15]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.14 to 0.24]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.86 to -0.37]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.18 to -0.01]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (CHA2DS2Vasc); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.64 to -0.21]

9. Primary Outcome: Number of Participants by Comedications
Description: Comedication was defined as the second or alternative medication used to relieve the side-effects of another medicine.
Time Frame: Up to 30 days after date of first prescription
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 4712 | 1423 | 32212 | 192 | 2286 | 363 | 2855 | 953 | 5132 | 1562
Participants | 4712 | 1406 | 32212 | 188 | 2286 | 352 | 2855 | 947 | 5132 | 1532
Statistical Analysis 1: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.008, Chi-squared; Odds Ratio (OR) = 1.88, 95% CI 2-sided [0.77 to 5.30]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.008, Chi-squared; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.33 to 1.12]
Statistical Analysis 3: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.008, Chi-squared; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.20 to 1.99]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants; Test type: Superiority; p = 0.008, Chi-squared; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.18 to 0.86]

10. Primary Outcome: Number of Participants With Apixaban Adherence With VKA, Dabigatran and Rivaroxaban as Assessed by Medication Possession Ratio (MPR)
Description: MPR was one of the methods of measuring adherence and was defined as the ratio of all days supply to elapsed days, during the 12-month observation period. All days supply defined as sum of number of days supply between the start date and last prescription dispensed. Elapsed days defined as number of days between the start date and the last prescription dispensed. There were three categories of adherence: poor defined as <80% of MPR, good defined as between 80% and 120% of MPR and over adherence defined as >120% of MPR.
Time Frame: Up to 12 months after date of first prescription
Population: Study population included all participants with a first-recorded prescription of apixaban, VKA, dabigatran or rivaroxaban for SPAF registered in SIDIAP database during the study and diagnosed with NVAF. Here "N" signifies number of participants evaluable for the specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 424 | 430 | 6108 | 32 | 344 | 79 | 447 | 311 | 527 | 495
Participants
  MPR: Poor adherence | 162 | 151 | 5634 | 31 | 103 | 57 | 241 | 177 | 147 | 131
  MPR: Good adherence | 259 | 276 | 460 | 0 | 151 | 13 | 206 | 133 | 378 | 360
  MPR: Over adherence | 3 | 3 | 14 | 1 | 90 | 9 | 0 | 1 | 2 | 4
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.14 to 1.75]
Statistical Analysis 2: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.67, 95% CI 2-sided [0.55 to 0.82]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.03 to 2.01]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.58, 95% CI 2-sided [1.23 to 2.04]
Statistical Analysis 5: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.44, 95% CI 2-sided [0.34 to 0.57]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.43, 95% CI 2-sided [0.02 to 3.73]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.52 to 0.84]
Statistical Analysis 8: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.95 to 1.36]
Statistical Analysis 9: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.06 to 3.41]
Statistical Analysis 10: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.65, 95% CI 2-sided [0.50 to 0.85]
Statistical Analysis 11: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.90 to 1.37]
Statistical Analysis 12: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.22 to 5.85]
Statistical Analysis 13: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 3.37, 95% CI 2-sided [2.86 to 3.99]
Statistical Analysis 14: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.11, 95% CI 2-sided [0.09 to 0.13]
Statistical Analysis 15: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.11 to 1.52]
Statistical Analysis 16: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.78 to 1.91]
Statistical Analysis 17: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.01, 95% CI 2-sided [0.00 to 0.09]
Statistical Analysis 18: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 2.07, 95% CI 2-sided [0.07 to 18.00]
Statistical Analysis 19: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.58, 95% CI 2-sided [0.45 to 0.75]
Statistical Analysis 20: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.41 to 0.63]
Statistical Analysis 21: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 29.40, 95% CI 2-sided [11.01 to 123.80]
Statistical Analysis 22: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Poor adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.91 to 1.86]
Statistical Analysis 23: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Good adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.10, 95% CI 2-sided [0.05 to 0.17]
Statistical Analysis 24: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Over adherence); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 9.73, 95% CI 2-sided [2.81 to 46.50]

11. Primary Outcome: Number of Participants With Apixaban Adherence With VKA, Dabigatran and Rivaroxaban as Assessed by Discontinuation Throughout the Year
Description: Discontinuation rate was defined as the lack of subsequent prescription of the index drugs within 2 months after last supply day of the last prescription. It was analyzed by calculating the treatment withdrawal or switch rate.
Time Frame: Up to 12 months after date of first prescription
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 1305 | 666 | 17434 | 117 | 1353 | 206 | 1449 | 559 | 1718 | 817
Participants | 881 | 236 | 11326 | 85 | 1009 | 127 | 1002 | 248 | 1191 | 322
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.92 to 1.27]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.15 to 1.83]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.93 to 1.27]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.96 to 1.47]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.79 to 1.01]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 4.82, 95% CI 2-sided [3.14 to 7.55]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 1.41, 95% CI 2-sided [1.19 to 1.67]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (Discontinuation first year); Test type: Superiority; p = 0.000, Chi-squared; Odds Ratio (OR) = 2.92, 95% CI 2-sided [2.12 to 4.05]

12. Primary Outcome: Apixaban Adherence With VKA, Dabigatran and Rivaroxaban by Number of Defined Daily Dose (NDDD)
Description: NDDD was a measure that represented the average daily maintenance dose for the main indication of a drug.
Time Frame: Up to 12 months after date of first prescription
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: milligrams per day
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
Number analyzed (Participants) | 1305 | 666 | 17434 | 117 | 1353 | 206 | 1449 | 559 | 1718 | 817
milligrams per day | 15.0 [15.0 to 30.0] | 30.0 [15.0 to 30.0] | 16.0 [16.0 to 32.0] | 16.0 [16.0 to 32.0] | 53.0 [53.0 to 53.0] | 16.0 [5.0 to 53.0] | 22.0 [22.0 to 29.0] | 22.0 [22.0 to 29.0] | 21.0 [15.0 to 28.0] | 28.0 [21.0 to 28.0]
Statistical Analysis 1: Comparison: Apixaban: Naive vs Dabigatran: Naive; Dabigatran vs. Apixaban in naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 3.63, 95% CI 2-sided [3.02 to 4.24]
Statistical Analysis 2: Comparison: Apixaban: Non Naive vs Dabigatran: Non-Naive; Dabigatran vs. Apixaban in non-naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.77 to 0.98]
Statistical Analysis 3: Comparison: Apixaban: Naive vs Rivaroxaban: Naive; Rivaroxaban vs. Apixaban in naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [0.84 to 2.17]
Statistical Analysis 4: Comparison: Apixaban: Non Naive vs Rivaroxaban: Non-Naive; Rivaroxaban vs. Apixaban in non-naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 1.98, 95% CI 2-sided [1.16 to 2.80]
Statistical Analysis 5: Comparison: Apixaban: Naive vs Acenocoumarol: Naive; Acenocumarol vs. Apixaban in naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.41 to 1.39]
Statistical Analysis 6: Comparison: Apixaban: Non Naive vs Acenocoumarol: Non-Naive; Acenocumarol vs. Apixaban in non-naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = -2.25, 95% CI 2-sided [-4.32 to -0.18]
Statistical Analysis 7: Comparison: Apixaban: Naive vs Warfarin: Naive; Warfarin vs. Apixaban in naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 28.52, 95% CI 2-sided [27.56 to 29.48]
Statistical Analysis 8: Comparison: Apixaban: Non Naive vs Warfarin: Non-Naive; Warfarin vs. Apixaban in non-naive participants (NDDDs); Test type: Superiority; p = 0.000, ANOVA; Mean Difference (Final Values) = 1.93, 95% CI 2-sided [-1.05 to 4.90]

13. Primary Outcome: International Normalized Ratio (INR) Values During the Last 12 Months Values in Participants Previously Treated With VKA
Description: INR was defined as the ratio of the participant's prothrombin time and the normal mean prothrombin time. Prothrombin time defined as a time taken by the blood to clot in participants receiving oral anticoagulant medication. INR was categorized according to the risk level: risk for coagulation (INR<2); optimal range (2<INR<3); and risk of hemorrhages (INR>3).
Time Frame: Up to 12 months after date of first prescription
Population: Study population included all participants with a first-recorded prescription of VKA for SPAF registered in SIDIAP database during the study and diagnosed with NVAF. Here "N" signifies number of participants evaluable for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive
Number analyzed (Participants) | 19192 | 113 | 872 | 158
ratio | 2.5 (0.4) | 2.5 (0.4) | 2.5 (0.3) | 2.6 (0.4)

14. Primary Outcome: Time in Therapeutic Range (TTR) Values During the Last 12 Months Values in Participants Previously Treated With VKA
Description: TTR was defined as the duration of time in which the participant's INR values were within a desired range (2 to 3). INR was defined as the ratio of the participant's prothrombin time and the normal mean prothrombin time. Prothrombin time defined as a time taken by the blood to clot in participants receiving oral anticoagulant medication. INR was categorized according to the risk level: risk for coagulation (INR<2); optimal range (2<INR<3); and risk of hemorrhages (INR>3).
Time Frame: Up to 12 months after date of first prescription
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non-Naive
Number analyzed (Participants) | 19192 | 113 | 872 | 158
days | 60.2 [47.2 to 71.8] | 59.6 [47.7 to 68.4] | 66.2 [52.2 to 77.4] | 58.9 [43.2 to 68.2]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected during the study
Description: Safety data was not planned to be collected during the study.
Arm/Group | Apixaban: Naive | Apixaban: Non Naive | Acenocoumarol: Naive | Acenocoumarol: Non-Naive | Warfarin: Naive | Warfarin: Non Naive | Dabigatran: Naive | Dabigatran: Non-Naive | Rivaroxaban: Naive | Rivaroxaban: Non-Naive
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03441633/Prot_SAP_000.pdf